CLINICAL TRIAL: NCT06898749
Title: Impact of Canine Mediation Practice in Psychomotor Therapy on Improving the Quality of Life in Adult Epileptic Patients.
Acronym: MCP-Epi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMR_2024_8
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- canine mediation in psychomotor therapy (Experimental): Group psychomotor therapy sessions combined with canine mediation
  (1 session per week for 10 weeks)
  Interventions: Other: canine mediation
- standard psychomotor therapy (Active Comparator): Standard group psychomotor therapy sessions (1 session per week for 10 weeks)
  Interventions: Other: standard psychomotor therapy

INTERVENTIONS:
Other: canine mediation — Animal mediation consists of bringing an animal into contact with a specific audience to improve the mental or physical health of a person. The dog and beneficiaries interact through various activities, in which the animal participates, offered during the sessions. The dog plays a particularly important role as a mediator through the bonds it forms with the human, as well as a non-judgmental partner in interaction.
  The canine educator will be accompanied by a healthcare professional during interventions. The sessions are organized based on the expertise and suggestions of both professions (canine educator and psychomotor therapist).
  The canine educator will be a state-certified professional educator with a specialization in animal mediation.
  The dog used is trained by the educator, with two types of learning being worked on: emotions and "commands" on cue.
  Arms: canine mediation in psychomotor therapy
Other: standard psychomotor therapy — standard sessions of psychomotor therapy
  Arms: standard psychomotor therapy

SUMMARY:
In addition to the search for new pharmaceutical or surgical solutions that could improve the therapeutic management of epileptic individuals, it is interesting to ask whether other complementary approaches, such as canine mediation in psychomotor therapy, could enhance the quality of life in this population.

However, there is currently no evidence indicating that exposure to animals through mediation sessions would be beneficial for epileptic individuals, particularly regarding their quality of life, anxiety, emotional management, or cognition (such as social cognition). In the absence of current data in this population, it seems pertinent to study the impact of this practice on people with epilepsy. Furthermore, beyond quality of life, it would be valuable to examine whether it also influences anxiety or the frequency of seizures in individuals with epilepsy (a phenomenon reported for epileptic individuals living with a pet dog or a service dog). Canine mediation could help better manage and regulate the emotions of epileptic individuals, as well as improve their self-esteem.

ELIGIBILITY:
Inclusion Criteria:

* Person aged ≥ 18 years
* Presenting pharmacoresistant epilepsy according to the criteria of the International League Against Epilepsy
* Requiring psychomotor therapy sessions for one of the following indications:

Difficult emotional and relational management And/or global motor difficulties And/or body schema organization disorder And/or temporo-spatial disorder

* Explicit consent or no opposition to participation in the study by the patient and/or their legal representative or guardian
* Image rights consented by the patient and their legal representative or guardian, if applicable
* Hospitalization or residence at the Teppe Institute or at the FAM (Foyer d'Accueil Médicalisé) des 4 Jardins planned for at least 3 months
* Affiliated with or a beneficiary of a social security scheme

Exclusion Criteria:

* Fear or phobia of dogs
* Epileptic person benefiting from a legal protection measure other than guardianship or curatorship
* Person with insufficient cognitive abilities to respond to the questionnaires
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of quality of life | Day 0 and Day 7 after the end of the 10 sessions
  Increase in the Quality of Life in Epilepsy Inventory-31 (QOLIE-31) score of at least 5 points between inclusion and one week after the completion of the 10 sessions.
  The score of the QOLIE-31 (Quality of Life in Epilepsy Inventory-31) ranges from 0 to 100. A score of 0 represents the worst possible quality of life, while a score of 100 represents the best possible quality of life.